CLINICAL TRIAL: NCT03483285
Title: Videolaryngoscopes in Open Heart Surgery
Brief Title: Comparison of Two Different Videolaryngoscopes Regarding Hemodynamic Parameters in Open Heart Surgey
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Tülay Çardaközü, Associate Professor, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: KOU-KAEK 2017-405
Record Dates: First submitted 2018-03-15; First posted 2018-03-30 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Intubation;Difficult; Coronary Bypass
Keywords: intubation; airtraq; open heart surgery; hemodynamic parameters

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- heart rate (Active Comparator): Effects of İntubation with Airtraq or Storz to heart rate
  Interventions: Device: airtraq; Device: storz
- mean arterial pressure (Active Comparator): Effect of intubation with Airtraq or Storz to mean arterial pressure
  Interventions: Device: airtraq; Device: storz

INTERVENTIONS:
Device: airtraq — airtraq videolaryngoscope
Device: storz — storz videolaryngoscope

SUMMARY:
Endotracheal intubation increased the heart rate and blood pressure in normal patients. Open heart surgery patients are more prone to hemodynamic variability. In addition, they have increased possibility for difficult intubation The heart rate and blood pressure increase impaired the oxygen consumption. This was previously shown that Videolaryngoscopes minimaly effects the vital signs in normal patients. Videolaryngoscopy inreased the rate of success in normal and difficult airway. This study aimed to compare two laryngoscopes regarding hemodynamic parameters and intubation times in coronary bypass surgery.

DETAILED DESCRIPTION:
Aim: Endotracheal intubation increased the heart rate and blood pressure in normal patients. Open heart surgery patients are more prone to hemodynamic variability. In addition, they have increased possibility for difficult intubation The heart rate and blood pressure increase impaired the oxygen consumption. This was previously shown that Videolaryngoscopes minimaly effects the vital signs in normal patients. Videolaryngoscopy inreased the rate of success in normal and difficult airway. This study aimed to compare two laryngoscopes regarding hemodynamic parameters and intubation times in coronary bypass surgery.

Material and methods: 50 patients undergoing coronary bypass surgery enrolled in this prospective.randomized study. Demogaphic variables and airway characteristics of patients were recorded. Glottic visulisation and intubation time were recorded. Systolic blood pressure, diastolic blood pressure, mean arterial pressure and heart rate were recorded 2 minutes intervals before intubation, after intubation during 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing open heart surgery
* < 18 years of age

Exclusion Criteria:

* emergency

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-21 (Actual)

PRIMARY OUTCOMES:
heart rate | 2 months
  heart rate

SECONDARY OUTCOMES:
insertion time | 2 months
  optimal glottic visualisation time
intubation time | 2 months
  intubation time
mean arterial pressure | 2 months
  mean arterial pressure

CONTACTS AND LOCATIONS:
Overall Officials: Tulay Cardakozu, Principal Investigator — Anesthesiology and Reanimation
Locations (1):
- Kocaeli University Hospital, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided